CLINICAL TRIAL: NCT02000804
Title: A Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of 160 mg Enteric-coated Micronised Free Base Darapladib in Healthy Chinese Subjects.
Brief Title: Darapladib China PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117326
Record Dates: First submitted 2013-06-20; First posted 2013-12-04 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Atherosclerosis
Keywords: Darapladib, Safety, Pharmacokinetics, Pharmacodynamics, Healthy Chinese Subjects
MeSH Terms: conditions — Atherosclerosis | interventions — darapladib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- darapladib 160mg (Experimental): drug
  Interventions: Drug: darapladib 160mg

INTERVENTIONS:
Drug: darapladib 160mg — drug

SUMMARY:
This study is to evaluate pharmacokinetics (PK), pharmacodynamics (PD) and safety of 160 mg enteric-coated micronised free base darapladib in healthy Chinese subjects.

DETAILED DESCRIPTION:
SB-480848 (darapladib) is a novel selective and orally active inhibitor of lipoprotein-associated phospholipase A2 (Lp-PLA2) being developed by GlaxoSmithKline (GSK) for the treatment of atherosclerosis.

This will be an open label study where each Subject will participate in 2 study sessions, a single dose session and a repeat dose session. All Subjects will receive 160 mg of enteric coated micronised free-base darapladib as a single dose and as repeated daily doses for 28 days.

The purpose of this study is to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) and safety of single and repeat oral dose of darapladib in healthy Chinese Subjects. The primary endpoints for safety are: clinical safety data from spontaneous adverse event reporting, 12-lead electrocardiogram recording, vital sign measurement, nursing/physician observation and clinical laboratory tests. The primary PK parameters of interest are area under plasma concentration time curve (AUC) and maximum plasma concentration (Cmax) of darapladib, while the secondary PK parameters of interest are: time of occurrence of Cmax (Tmax) and apparent terminal phase half-life (t1/2) of darapladib as well as AUC, Cmax, Tmax and t1/2 of the metabolite, SB-553253. Finally, the PD endpoint of interest is plasma Lp PLA2 activity, as expressed in terms of percent inhibition relative to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese males or females aged between 18 and 45 years of age inclusive, at the time of signing the informed consent. (Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A Subject with a clinical abnormality or laboratory parameters which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator (in consultation with the GSK Medical Monitor if required) agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. )
* Of Chinese origin - defined as being born in mainland China, having four ethnic Chinese grandparents.
* Body weight ≥50 kg and BMI within the range 19 to 24 kg/m2 (inclusive).
* A female Subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the Subject's medical history for study eligibility, as obtained via a verbal interview with the Subject or from the Subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory].

Child-bearing potential with negative pregnancy test as determined by urine human chorionic gonadotropin (hCG) test at screening or prior to dosing and Agrees to use 1 of the contraception methods listed in Section 4.3.1 from the time of Screening to sufficiently minimize the risk of pregnancy at that point. Female Subjects must agree to use contraception until the follow-up contact.

* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Alanine aminotransferase (ALT), alkaline phosphatise (ALP) and bilirubin ≤1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Based on single or averaged QTc values of triplicate ECGs obtained over a brief recording period:

QT duration corrected for heart rate by Bazett's formula (QTcB) or QT duration corrected for heart rate by Fridericia's formula (QTcF) <450 msec; QTc <480 msec in Subjects with Bundle Branch Block.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Consumption of grapefruit or grapefruit juice within 7 days prior to first dose of study medication.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of asthma, anaphylaxis or anaphylactoid reactions, severe allergic responses.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* A positive test for Hepatitis B surface antigen (HBsAg) or positive Hepatitis C antibody result, or positive test for human immunodeficiency virus (HIV) antibody or Syphilis antibody at Screening.
* A positive pre-study drug/alcohol screen.
* Pregnant females as determined by positive urine hCG test at screening or prior to dosing.
* A chest X-ray or computed tomography (CT) scan that reveals evidence of clinical significant abnormalities eg, tuberculosis. A chest X-ray must be taken at Day-1 if a chest X-ray or CT scan is not available within 6 months prior to that day.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The Subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10-23 (Actual); Primary Completion 2014-01-04 (Actual); Study Completion 2014-01-04 (Actual)

PRIMARY OUTCOMES:
Adverse event | Up to 12 weeks
  An AE is any untoward medical occurrence in a patient or clinical investigation Subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
12-lead ECG | Up to 12 weeks
  12-lead ECGs will be obtained at designated timepoint during the study, using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTc intervals.
Vital sign measurement | Up to 12 weeks
  Systolic and diastolic blood pressure and pulse rate
clinical laboratory examination | Up to 12 weeks
  Hematology, clinical chemistry, urinalysis and additional parameters to be tested
AUC0-t for darapladib | Up to 12 weeks
  Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration
AUC 0-∞ for Darapdlib | Up to 12 weeks
  Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time
Cmax for darapladib | Up to 12 weeks
  Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time
Rcmax for darapladib | Up to 12 weeks
  Accumulation ratios Cmax accumulation ratio
Ro for darapladib | Up to 12 weeks
  Accumulation ratios Cmax accumulation ratio
Nursing/physician observation | Up to 12 weeks
  The physical examination will include assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen).

SECONDARY OUTCOMES:
Tmax for darapladib | Up to 12 weeks
  Time of occurrence of Cmax for darapladib
T1/2 for darapladib | Up to 12 weeks
  Terminal phase half-life for darapladib
AUC0-t for darapladib metabolite SB-553253 (as data permit). | Up to 12 weeks
  Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration for the pharmacologically active metabolite SB-553253
AUC0-∞ for darapladib metabolite SB-553253 (as data permit). | Up to 12 weeks
  Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time the pharmacologically active metabolite SB-553253
Cmax for darapladib metabolite SB-553253 (as data permit). | Up to 12 weeks
  Maximum observed concentration for the pharmacologically active metabolite SB-553253
T1/2 for darapladib metabolite SB-553253 (as data permit). | Up to 12 weeks
  Terminal phase half-life for the pharmacologically active metabolite SB-553253
Tmax for darapladib metabolite SB-553253 (as data permit). | Up to 12 weeks
  Time of occurrence of Cmax for the pharmacologically active metabolite SB-553253
Plasma Lp-PLA2 activity | Up to 12 weeks
  Percent inhibition relative to baseline of Plasma Lp-PLA2

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Hu C, Tompson D, Magee M, Chen Q, Liu YM, Zhu W, Zhao H, Gross AS, Liu Y. Single and Multiple Dose Pharmacokinetics, Pharmacodynamics and Safety of the Novel Lipoprotein-Associated Phospholipase A2 Enzyme Inhibitor Darapladib in Healthy Chinese Subjects: An Open Label Phase-1 Clinical Trial. PLoS One. 2015 Oct 14;10(10):e0139862. doi: 10.1371/journal.pone.0139862. eCollection 2015. PMID 26465780
- See also: Results for study 117326 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/117326?search=study&study_ids=117326#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 117326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117326 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register